CLINICAL TRIAL: NCT04443218
Title: Edwards PASCAL Transcatheter Valve Repair System Registry: A Multicenter Observational Registry With the Edwards PASCAL Transcatheter Valve Repair System
Brief Title: Edwards PASCAL Transcatheter Valve Repair System Registry
Acronym: PASCALRegistry
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-03
Record Dates: First submitted 2020-04-01; First posted 2020-06-23 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Edwards PASCAL Transcatheter Valve Repair System — The Edwards PASCAL Valve Repair System is indicated for the percutaneous reconstruction of an insufficient mitral valve.

SUMMARY:
This registry will collect prospective and retrospective clinical data on patients treated with the Edwards PASCAL Transcatheter Valve Repair System outside of the Post-Market Clinical Follow-up (PMCF) study.

DETAILED DESCRIPTION:
Patients treated per standard of care at their medical facilities and a written informed consent will be collected to allow the data to be collected. This registry intends to enroll patients under commercial usage and will serve as a mechanism to collect clinical data to further characterize the safety, performance and effectiveness of the PASCAL Transcatheter Valve Repair System.

ELIGIBILITY:
Inclusion Criteria:

* Patient signs informed consent to participate in the registry
* Patient is intended to or has received the PASCAL device

Exclusion Criteria:

* Patient does not consent to participate
* Patient is part of an ongoing Edwards Pre or Post Market Clinical study for the PASCAL Transcatheter Valve Repair System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Mitral Regurgitation eligible to receive the PASCAL device
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Hausleiter, Prof., Principal Investigator — MD
Locations (14):
- Germany (13):
  - LMU Klinikum der Universität München, München, Bavaria
  - Immanuel Klinikum Bernau, Bernau bei Berlin, Brandenburg
  - Universitätsklinikum Gießen, Giessen, Hesse
  - Georg-August-Universität Göttingen, Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - Herzzentrum Köln, Cologne, Nord Rhine Westphalia
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen, North Rhine-Westphalia
  - Herzzentrum der Universitätsklinik Bonn, Bonn, North Rhine-Westphalia
  - St.-Johannes-Hospital Dortmund, Dortmund, North Rhine-Westphalia
  - Elisabeth-Krankenhaus Essen, Essen, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Herzzentrum Universitätsklinik Dresden, Dresden, Saxony
  - Heart Centre of the University Leipzig, Leipzig, Saxony
  - Kath. Marienkrankenhaus Hamburg GmbH, Hamburg
- Inselspital Bern, Bern, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- Edwards PASCAL Transcatheter Mitral Valve Repair System: Mitral valve repair with PASCAL implanted via transcatheter procedure
Period: Overall Study
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Started | 220
Completed | 187
Not Completed | 33
Not completed — Exited study for other reasons | 9
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 4
Not completed — Death | 19

BASELINE CHARACTERISTICS:
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.2 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 138
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Data unavailable for 2 patients
  kg/m^2
    number analyzed (Participants) | 218
    (all) | 26.2 (5.15)
STS Score for Mitral Valve Repair [Mean (Standard Deviation); unit: %] — The Society of Thoracic Surgeons (STS) Score for Mitral Valve Repair is a validated risk-prediction model for operative mortality associated with mitral valve repair surgery based on the STS Adult Cardiac Care Surgery Database. In general, an STS predicted risk score of 4%-8% is considered intermediate risk and 8% or greater is considered high risk Population: Data unavailable for 62 patients
  %
    number analyzed (Participants) | 158
    (all) | 4.1 (3.11)
EuroScore II [Mean (Standard Deviation); unit: %] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) II is a cardiac risk model for predicting mortality after cardiac surgery. The higher the score, the higher the risk of an adverse outcome
  EuroScore II risk levels are as follows:
  Low risk: <8% Moderate risk: 8-10% High risk: >10% Population: Data unavailable for 17 patients
  %
    number analyzed (Participants) | 203
    (all) | 7.6 (8.20)
New York Heart Association (NYHA) Functional Class [Count of Participants; unit: Participants] — NYHA Functional Classification is a 4-category system commonly used by physicians to assess patient heart failure symptoms based on limitations to physical activity:
  Class I - No symptoms and no limitation in ordinary physical activity. Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Population: Data unavailable for 4 patients
  Participants
    number analyzed (Participants) | 216
    Class I | 3
    Class II | 33
    Class III | 161
    Class IV | 19
Mitral Regurgitation (MR) Etiology [Count of Participants; unit: Participants] — Underlying cause of MR, includes functional, degenerative, mixed (both functional and degenerative), and other Population: Data unavailable for 2 patients
  Participants
    number analyzed (Participants) | 218
    Functional MR | 106
    Degenerative MR | 85
    Mixed MR | 23
    Other | 4
Mitral Regurgitation (MR) Severity [Count of Participants; unit: Participants] — MR severity was assessed by sites using a 5-grade scale: none/trace (0-1+), mild (1+), mild to moderate (2+), moderate to severe (3+), and severe (4+).
  Participants
    None/Trace (0-1+) | 0
    Mild (1+) | 0
    Mild to Moderate (2+) | 1
    Moderate to Severe (3+) | 137
    Severe (4+) | 82

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Events (MAEs)
Description: Composite rate of all-cause death, myocardial infarction, stroke, heart failure hospitalization, or complication requiring transcatheter or surgical intervention (repeat transcatheter edge-to-edge repair [TEER] or mitral valve surgery)
Time Frame: 30 days
Population: Analysis includes patients who had an MAE or who were followed for at least 30 days. Patients may experience more than one MAE.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 216
Participants
  Composite MAE | 9
  All-cause death | 2
  Myocardial infarction | 0
  Stroke | 1
  Heart failure hospitalization | 5
  Complication requiring transcatheter or surgical intervention (repeat TEER or mitral valve surgery) | 2

2. Primary Outcome: Mitral Regurgitation (MR) Reduction to <=2+
Description: MR severity assessed by sites using a 5-grade scale: none/trace (0-1+), mild (1+), mild to moderate (2+), moderate to severe (3+), and severe (4+).
Time Frame: 30 days, 12 months
Population: Outcome data collected per standard of care at each investigative site and analyzed, if available. Analysis population includes participants with available data at one or more timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 191
Participants
  30 days: number analyzed (Participants) | 163
  30 days | 155
  12 months: number analyzed (Participants) | 133
  12 months | 122

3. Secondary Outcome: Quality of Life, as Assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Scores
Description: KCCQ is a 23-item, self-administered, validated questionnaire that quantifies physical function, symptoms, social function, self-efficacy, and quality of life for patients with heart failure. Scores range from 0 to 100 with higher scores indicating better function (100 = no symptoms, no limitations, and excellent quality of life).
Time Frame: Baseline, 30 days, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 107
Score on a scale
  Baseline: number analyzed (Participants) | 65
  Baseline | 45.3 (19.93)
  30 Days: number analyzed (Participants) | 55
  30 Days | 59.1 (20.89)
  12 Months: number analyzed (Participants) | 70
  12 Months | 71.0 (21.83)

4. Secondary Outcome: Quality of Life, as Assessed by EQ-5D Visual Analog Scale (VAS)
Description: Patient's self-rated health on a visual analog scale (0-100 points; 0=worst health you can imagine and 100=best health you can imagine).
Time Frame: Baseline, 30 days, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 85
Score on a scale
  Baseline: number analyzed (Participants) | 39
  Baseline | 51.9 (18.16)
  30 Days: number analyzed (Participants) | 40
  30 Days | 60.6 (17.77)
  12 Months: number analyzed (Participants) | 55
  12 Months | 61.6 (20.21)

5. Secondary Outcome: New York Heart Association (NYHA) Functional Classification
Description: NYHA Functional Classification is a 4-category system commonly used by physicians to assess patient heart failure symptoms based on limitations to physical activity:
  Class I - No symptoms and no limitation in ordinary physical activity. Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest.
Time Frame: Baseline, 30 days, 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 220
Participants
  Baseline: number analyzed (Participants) | 216
  Baseline: Class I | 3
  Baseline: Class II | 33
  Baseline: Class III | 161
  Baseline: Class IV | 19
  30 Days: number analyzed (Participants) | 183
  30 Days: Class I | 29
  30 Days: Class II | 89
  30 Days: Class III | 64
  30 Days: Class IV | 1
  12 Months: number analyzed (Participants) | 169
  12 Months: Class I | 28
  12 Months: Class II | 73
  12 Months: Class III | 67
  12 Months: Class IV | 1

6. Secondary Outcome: 6-Minute Walk Test (6MWT)
Description: 6MWT is a submaximal exercise test that measures the distance that a patient can walk on a flat surface in a period of 6 minutes.
Time Frame: Baseline, 30 days, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 119
meter
  Baseline: number analyzed (Participants) | 83
  Baseline | 275.5 (116.16)
  30 Days: number analyzed (Participants) | 78
  30 Days | 292.9 (119.92)
  12 Months: number analyzed (Participants) | 59
  12 Months | 310.2 (108.30)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
All-Cause Mortality (participants affected / at risk) | 19/220
Serious Adverse Events (participants affected / at risk) | 82/220
Other Adverse Events (participants affected / at risk) | 0/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards PASCAL Transcatheter Mitral Valve Repair System (N=220)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Readmission - Cardiac (not Heart Failure) (Cardiac disorders) | 26 (30)
Readmission - Heart Failure (Cardiac disorders) | 35 (51)
Atrial Septal Defect (ASD) Closure Due to Transseptal Catheterizaton (Injury, poisoning and procedural complications) | 2 (2)
Bleeding at Access Site (Injury, poisoning and procedural complications) | 1 (1)
Hematoma at Access Site (Injury, poisoning and procedural complications) | 1 (1)
Major Vascular Complication (Injury, poisoning and procedural complications) | 1 (1)
Other Device Related Event (Product Issues) | 3 (3) — Includes but is not limited to Single Leaflet Device Attachment events that occurred during follow-up.
Single Leaflet Device Attachment (Product Issues) | 1 (1) — Includes Single Leaflet Device Attachment events reported during procedure visit only. Single Leaflet Device Attachment events occurring during follow-up reported as Other Device Related Event.
New Requirement for Dialysis (Renal and urinary disorders) | 4 (6)
Complication Requiring Transcatheter or Surgical Intervention (Surgical and medical procedures) | 2 (2)
Mitral Valve Re-Intervention (Surgical and medical procedures) | 4 (5)
Readmission - Non-Cardiac (Follow Up) (Surgical and medical procedures) | 22 (30)
Unplanned Other Cardiac Surgery or Intervention (Not Mitral Valve Re-Intervention) (Surgical and medical procedures) | 16 (27)
Unplanned Vascular Surgery or Intervention (for Bleeding or Access Site Complication) (Surgical and medical procedures) | 1 (1)
Life-Threatening Bleeding (Vascular disorders) | 1 (2)
Major Bleeding Event (Vascular disorders) | 3 (3)
Other Bleed (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Interpretation of some outcome measures is limited by significant incomplete and/or missing data due to retrospective data collection, differences in data collected as part of standard of care across sites, and use of alternative follow-up data collection methods in lieu of in-person clinical visits. Additionally, this registry did not use an echocardiography core laboratory to assess echocardiography parameters or a clinical events committee to adjudicate adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication or presentation of the overall registry results and/or site-specific results requires prior written approval of Edwards.

DOCUMENTS (2):
  • Study Protocol (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT04443218/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT04443218/SAP_001.pdf